CLINICAL TRIAL: NCT04487938
Title: THE HONG KONG ORAL CANCER EDUCATION AND SCREENING (HOCES) PROGRAM: REFINING DISEASE PREVENTION, RISK STRATIFICATION AND EARLY DETECTION
Brief Title: Oral Cancer Screening and Education in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Peter James Thomson, Professor, The University of Hong Kong
Other Study IDs: thomsonp@hku.hk
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Oral Cancer; Oral Leukoplakia; Oral Submucous Fibrosis; Proliferative Verrucous Leukoplakia; Oral Erythroplakia; Erosive Lichen Planus
MeSH Terms: conditions — Mouth Neoplasms; Leukoplakia, Oral; Oral Submucous Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral rinse samples obtained via drooling in 50cc tubes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tobacco use and/or alcohol consumption
  Interventions: Other: No intervention utilised
- No tobacco use and/or alcohol consumption
  Interventions: Other: No intervention utilised

INTERVENTIONS:
Other: No intervention utilised — No intervention utilised

SUMMARY:
This study will be conducted to obtain data on oral cancer risk factors to generate machine learning models with good predictive accuracy for stratifying individuals with high-oral cancer risk and delineating high-risk and low-risk oral lesions. Likewise, this study will seek to provide oral cancer-related health education and training on oral-self-examination for beneficiaries

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals satisfying age and residential area criteria with no previous history of oral cancer. Individuals with a history of other cancers will be included in the study provided they have been in remission for more than three years.

Exclusion Criteria:

* Participants with reduced mouth opening (irrespective of the cause) to permit proper administration of VOE or photosensitive epilepsy will be excluded. Likewise, those who decline the provision of written consent or participation in any part of the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hong Kong residents aged 45 years and above residing in Southern and Central and Western district council districts (DCD).
Sampling Method: Non-Probability Sample
Enrollment: 3190 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of machine learning algorithms for predicting high-risk persons | 24 months
  Predictive accuracy of the ML classifiers for forecasting individuals with or likely to develop high-risk lesions within 24 months of first screening encounter based on demographic and lifestyle information.
Accuracy of machine learning algorithms for discriminating high-risk and low-risk lesions | 24 months
  Predictive accuracy of ML classifiers for classifying high-risk and low-risk lesions based on demographic and lifestyle risk factors, oral high-risk HPV status, and salivary DNA hypermethylation levels.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Thomson, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adeoye J, Choi SW, Thomson P. Bayesian disease mapping and the 'High-Risk' oral cancer population in Hong Kong. J Oral Pathol Med. 2020 Oct;49(9):907-913. doi: 10.1111/jop.13045. Epub 2020 Jun 10. PMID 32450000
- [Background] Adeoye J, Brennan PA, Thomson P. "Search less, verify more"-Reviewing salivary biomarkers in oral cancer detection. J Oral Pathol Med. 2020 Sep;49(8):711-719. doi: 10.1111/jop.13003. Epub 2020 Mar 5. PMID 32027406
- [Background] Adeoye J, Chu CS, Choi SW, Thomson P. Oral Cancer Awareness and Individuals' Inclination to Its Screening and Risk Prediction in Hong Kong. J Cancer Educ. 2022 Apr;37(2):439-448. doi: 10.1007/s13187-020-01834-x. PMID 32705524
- [Background] Adeoye J, Thomson P. Strategies to improve diagnosis and risk assessment for oral cancer patients. Faculty Dental Journal. 2020;11(3):122-7.